CLINICAL TRIAL: NCT05005325
Title: Functional Movement Screen Differences in Male and Female Footballers as an Injury Prevention Tool.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REC/0867 Fatima Amjad
Record Dates: First submitted 2021-08-05; First posted 2021-08-13 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Sports Physical Therapy
Keywords: Functional Movement Screen,; Footballers,; Speed

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group(Male) (Active Comparator): Participants will be included in the study after screening from inclusion criteria. Each participant will perform FMS during a single session before competition as pre testing. It consists of 7 movement tasks and 3 clearance screens. Movement task will include deep squat, hurdle step, inline lunge, shoulder mobility, active straight-leg raise, trunk stability push-up and rotary stability. Five of the 7 tasks (hurdle step, inline lunge, shoulder mobility, active straight-leg raise and rotary stability) will be performed on both right and left sides. In addition to these, 3 clearance screen will assess the presence of pain with shoulder internal rotation/flexion, end range spinal flexion and end range spinal extension. Participants will be instructed for each task performance and will perform 3 attempts for each task.
  Interventions: Other: Experimental group(Male)
- Experimental group(Female) (Experimental): Participants will be included in the study after screening from inclusion criteria. Each participant will perform FMS during a single session before competition as pre testing. It consists of 7 movement tasks and 3 clearance screens. Movement task will include deep squat, hurdle step, inline lunge, shoulder mobility, active straight-leg raise, trunk stability push-up and rotary stability. Five of the 7 tasks (hurdle step, inline lunge, shoulder mobility, active straight-leg raise and rotary stability) will be performed on both right and left sides. In addition to these, 3 clearance screen will assess the presence of pain with shoulder internal rotation/flexion, end range spinal flexion and end range spinal extension. Participants will be instructed for each task performance and will perform 3 attempts for each task.
  Interventions: Other: Experimental group(Female)

INTERVENTIONS:
Other: Experimental group(Male) — Hurdle steps Deep squats Inline lunges Shoulder Clearing Active straight leg raise Trunk stability pushup Rotary stability Spinal extension exam Spinal flexion exam
  Arms: Experimental group(Male)
Other: Experimental group(Female) — Hurdle steps Deep squats Inline lunges Shoulder Clearing Active straight leg raise Trunk stability pushup Rotary stability Spinal extension exam Spinal flexion exam
  Arms: Experimental group(Female)

SUMMARY:
Football is definitely a sport commonly held across the world. It is played mostly at the professional level and as a leisure sport as well. Many countries organize football matches at different levels, and these matches include various age groups ranging from adolescents to young adults. As the participation in football is increasing it is also increasing the risk of developing injuries. It exposes the athlete to contact injuries and non-contact injuries. The intensity of the body's biomechanical and physiological reactions when playing football is enhanced because it has sporadic and irregular activity. This increased workload can increase the risk of injury. Many sport specialists perform movements which are related to that specific sport but the paradigm has been shifted to a more integrated functional approach which includes principles of proprioceptive neuromuscular facilitation, muscle synergy and motor learning and it is important to inspect the basic fundamental movements as these occur throughout many athletic activities. Before participating in the sporting event, athletes undergo a comprehensive pre-participation examination which includes examination of health status, underlying medical problems and musculoskeletal system, it is a standard approach to injury screening. However, this does not evaluate the intrinsic risk factors which might be associated with the injury during field.

DETAILED DESCRIPTION:
Functional movement screening (FMS) was developed by Cook et al. It evaluates range of motion, muscular imbalances and core strength by means of seven different movement. It is used to analyze the pattern of various fundamental movements and then highlights the limitations in that pattern and recognizes asymmetries in relation to that pattern of movement and eventually compares these inadequacies with outcomes that will improve a pragmatic approach to injury prevention. Prior studies reported that during pre-participation FMS can predict injuries in various athletes.

Several research studies carried out by researchers in this area have been involved in the exploring the strategies that can enhance the efficiency and performance of footballers in the field and investigate the effects of injuries on performance. Studies including FMS as an injury and evaluation tool have subjects which includes athletes playing multiple sports and generally involved male footballers, but the studies comparing scores of FMS among female footballers with male footballers are scarce. With advances in society and knowledge of participation in sports, more women participate in sports events, and the pre-participation and injury of this particular population should be explored. This research will discover this particular issue and bring to light the needs of female footballers and contributes to recognizing FMS as a predictive method for injury.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female Footballers
* Athletes training at least 3 times per week (>1.5h/week)

Exclusion Criteria:

* Recent injury of lower extremity within past 6 months
* History of traumatic brain injury
* History of concussion
* History of cervical spine injury within the last year
* History of shoulder surgery
* History of anterior cruciate ligament repair
* History of meniscal repair
* History of Achilles tendon repair
* History of ankle fracture
* Recent eye and ear disorders within past 6 months
* Receiving physical therapy for musculoskeletal injuries

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 264 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Functional Movement Screen | 6th week
  Functional Movement Screen (FMS) will be used as a 'Pre' and 'Post' assessment tool to evaluate the risk of injury/dysfunctional performance among male and female footballers.
  Minimum and Maximum score interpretation required

CONTACTS AND LOCATIONS:
Overall Officials: Danish Latif, MSPT-SPT, Principal Investigator — Riphah International University
Locations (1):
- Ra'ad Arena, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No